CLINICAL TRIAL: NCT01031108
Title: A Phase I, Randomized, Placebo-Controlled, Crossover Clinical Trial to Assess the Safety of Oral SRT2104 and Its Effects on Vascular Dysfunction in Otherwise Healthy Cigarette Smokers and Subjects With Type 2 Diabetes Mellitus
Brief Title: A Clinical Trial to Assess the Safety of Oral SRT2104 and Its Effects on Vascular Dysfunction in Otherwise Healthy Cigarette Smokers and Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 114089
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type 2 Diabetic Group (Other): The Type 2 Diabetic Treatment Group will be randomized to receive test material (2.0g SRT2104 or placebo) in the form of 8 capsules per day for 28 days. After 28 days of dosing, subjects will cross over to receive placebo or 2.0g SRT2104 for an additional 28 days. Dosing of SRT2104 or placebo will take place at approximately the same time every morning, approximately 15 minutes following consumption of a standardized morning meal (220 cc of Ensure Plus®). Subjects must wait at least 1-2 hours after dosing before consuming additional calories. Water is permitted ad libitum.
  Interventions: Drug: Placebo; Drug: SRT2104
- Otherwise Healthy Cigarette Smoking Group (Other): The Otherwise Healthy Cigarette Smoking Treatment Group will be randomized to receive test material (2.0g SRT2104 or placebo) in the form of 8 capsules per day for 28 days. After 28 days of dosing, subjects will cross over to receive placebo or 2.0g SRT2104 for an additional 28 days. Dosing of SRT2104 or placebo will take place at approximately the same time every morning, approximately 15 minutes following consumption of a standardized morning meal (220 cc of Ensure Plus®). Subjects must wait at least 1-2 hours after dosing before consuming additional calories. Water is permitted ad libitum.
  Interventions: Drug: Placebo; Drug: SRT2104

INTERVENTIONS:
Drug: Placebo — For the placebo product, SRT2104 drug substance will be replaced by microcrystalline cellulose (Avicel® PH 105) to match the SRT2104 investigational product.
  Eight placebo capsules are stored in a dosing bottle and provided to all participating subjects for oral ingestion.
Drug: SRT2104 — SRT2104 investigational product is a size 00 Swedish Orange opaque hard gelatin capsule containing 0.25 g of SRT2104, a new chemical entity which is supplied as a micronized, yellowish/amber powder. Eight SRT2104 capsules are stored in a dosing bottle and provided to all participating subjects for oral ingestion.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of SRT2104 (2.0 g administered once daily for 28 days) and to examine the effects of SRT2104 (2.0 g administered once daily for 28 days) on reversing vasomotor and fibrinolytic dysfunction in both type 2 diabetes mellitus patients and otherwise healthy cigarette smokers in a fed state.

This study will investigate the effects of SRT2104 on the reduction of platelet activation markers (platelet-monocyte aggregates), and to evaluate the effects of SRT2104 on platelet and monocyte surface markers (P-selectin, CD11b), inflammatory markers (high sensitivity CRP, IL-6, SAA, TNF-α and sCD40L), and markers of oxidative stress (urinary and plasma F2-isoprostanes and nitrotyrosine).

Further goals of this study is to characterize the pharmacokinetic profile of SRT2104 after a single dose and multiple administrations in both type 2 diabetes mellitus patients and otherwise healthy cigarette smokers in a fed state, and to explore the effects of SRT2104 on potential biomarkers of activity for glucose control (HbA1c, glycated albumin and fructosamine) and/or Sirt1 activation.

DETAILED DESCRIPTION:
Single-center, randomized, double-blind, placebo-controlled, crossover, safety, activity, and pharmacokinetic (PK) study of 2.0 g of SRT2104 administered orally once daily for 28 consecutive days to two different populations: type 2 diabetic (T2D) subjects on an existing, stable, hypoglycemic regimen and otherwise healthy cigarette smokers (≥ 10cigarettes/day for at least 1 year). Approximately 24 subjects with T2D and 24 otherwise healthy cigarette smokers, aged 18-60 years, who fulfill the inclusion/exclusion criteria, will be enrolled in this study to ensure at least 20 evaluable subjects per population are enrolled. Subjects will be evenly stratified and randomized to receive SRT2104 2.0 g/day or placebo once daily for 28 days. After 28 days, subjects will cross over to receive the other test article for another 28 days of dosing, bringing the total dosing period to 56 days.

Subjects will sign the informed consent form at the screening visit (to occur within 21 days of first dose of test article), and will undergo screening assessments to verify eligibility for the study. If eligible and willing to participate, subjects will return to the clinic on Days -1 and 1 for safety assessments, hematology and biochemistry measurements, platelet monocyte aggregation (PMA) assessment, forearm venous occlusion plethysmography, pulse wave analysis (PWA), pulse wave velocity (PWV) and PK sampling. The first dose of test article will occur on Day 1 after eligibility has been confirmed. After each 28 day dosing period, subjects will return on Day 28 and Day 56 for safety assessments, hematology and biochemistry measurements, forearm plethysmography, PWA, PWV, and PK sampling. Subjects will return to the clinic on Days 2, 15, 29, 43, and 57 for safety assessments and additional PK sampling. Subjects will be asked to complete a study drug diary on a daily basis for compliance and adverse event (AE) monitoring (diabetic subjects will be required to monitor and record their fasting blood glucose in the diary also). An End of Study visit will occur 14 days following the final dose of SRT2104 or placebo on Day 70. A followup safety call will be made to each subject 30 days following their final dose of SRT2104 or placebo (Day 86).

ELIGIBILITY:
Inclusion Criteria:

- Ambulatory male and female subjects (of any race) either with type 2 diabetes or otherwise healthy cigarette smokers (≥ 10 cigarettes/day for at least 1 year) within the age range of 18-70 years (inclusive) at the time of Screening.

* If a subject is diabetic, HbA1c at Screening is < 9.0%
* If a subject is diabetic, fasting plasma glucose (FPG) ≤ 13.875 mmol/L (≤ 250 mg/dL).
* If a subject is diabetic, an official diagnosis of type 2 diabetes must be documented for at least 6 months prior to first dose of test article.
* If a subject is diabetic, subject must be on an existing, stable, hypoglycemic therapy or a stable dietary regimen to control their disease for at least 3 months prior to Screening.

Note: If a subject is a diabetic and a smoker, then they are not eligible for the trial. A minimum 5 year non-smoking history is required for all type 2 diabetic subjects to be enrolled into the study.

* Female subjects of child-bearing potential, willing to use reliable contraception (see Section 5.10) for the duration of the study, through to the 30 day safety follow up visit (a female of child-bearing potential is defined as any female, regardless of her age with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility. Females with oligomenorrhea or who are perimenopausal, and young females who have begun to menstruate are considered to be of child-bearing potential)
* All male subjects must agree with their partners to use double-barrier birth control or abstinence while participating in the study and for 12 weeks following the last dose of study drug.
* Willingness to provide written informed consent to participate in the study.
* Subject may be on concomitant treatments for other conditions, provided the medical condition necessitating the treatment and therapy is stable for at least 3 months prior to screening and the treatment is not counterindicated by the study protocol.
* Subject is not currently on a therapeutic regimen of ACE inhibitors, anti-coagulants, anti-platelets, or any other medications or treatments which may influence coagulation (with the exception of 81 mg or less of aspirin/acetylsalicylic acid daily).
* Body Mass Index (BMI) of 18.5-38 kg/m^2 (inclusive).
* Resting supine blood pressure (BP) <160/90 mmHg.
* Absence of significant disease (other than type 2 diabetes) or clinically significant abnormal laboratory values on the laboratory evaluations, medical history, or physical examination during screening; normal end organ function at the discretion of the principal investigator.
* Negative test result at screening for HIV 1 and 2.
* Negative test result at screening for hepatitis B & C virus.
* Have a normal 12-lead electrocardiogram (ECG) or one with changes considered to be clinically insignificant on medical review. QTcB must be < 450 msec for males and females. QTcB must be <480 msec in subjects with Bundle Branch Block.
* Comprehension of the nature and purpose of the study and compliance with the requirements of the entire protocol.
* Able to communicate in person and by telephone in a manner that allows all protocol procedures to be carried out safety and reliably in the opinion of the investigative site staff.

Exclusion Criteria:

* If diabetic, any major illness in the past 3 months or any significant ongoing chronic medical illness not related to diabetes which in the opinion of the principal investigator or medical monitor could risk subject safety or interpretation of the results.
* If an otherwise healthy cigarette smoker, any major illness or injury in the past 3 months or any significant ongoing chronic medical illness (including diabetes) which in the opinion of the principal investigator or medical monitor could risk subject safety or interpretation of the results.
* Renal or liver impairment, defined as alkaline phosphatase and/or bilirubin ≥ 1.5 x ULN (an isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%), serum creatinine level of ≥ 123.76 µmol/L (≥ 1.4 mg/dL ) in females and ≥ 132.60 µmol/L (≥ 1.5 mg/dL ) in males, and > 2 × ULN for liver transaminases (ALT and AST), respectively.
* History of or current gastrointestinal diseases or surgeries influencing drug absorption, except for appendectomy.
* History, within 3 years, of drug abuse (including benzodiazepines, opioids, amphetamine, cocaine, and THC).
* History of alcoholism (more than 2 years), moderate drinkers (more than three drinks per day) or having consumed alcohol within 48 hours prior to first dose of test article (one drink is equal to one unit of alcohol [one glass wine, half pint beer, one measure of spirit]).
* Participation in any clinical trial within the past 3 months prior to the first dose of test article in the current study.
* History of difficulty in donating blood or accessibility of veins in left or right arm.
* Donation of blood or loss of blood (greater than 500 mL) within 3 months prior to receiving the first dose of test material.
* Use of any dietary or herbal supplements within 2 weeks prior the first dose of study drug, with the exception of an Investigator approved vitamin.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Active neoplastic disease or history of neoplastic disease within 5 years of study entry (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ).
* A positive pre-study drug screen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-05-28 (Actual); Primary Completion 2011-10-12 (Actual); Study Completion 2011-10-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of SRT2104 (2.0 g administered once daily for 28 days) in both type 2 diabetes mellitus patients and otherwise healthy cigarette smokers in a fed state. | AEs and clinically significant abnormal laboratory values will be recorded based upon investigator observation and subject reporting through a subject diary. Safety will be monitored by AEs, VS, physical exam, labs and ECGs during the study.
To examine the effects of SRT2104 (2.0 g administered once daily for 28 days) on reversing vasomotor and fibrinolytic dysfunction in both type 2 diabetes mellitus patients and otherwise healthy smokers in a fed state. | Forearm venous occlusion plethysmography will be performed on Days -1, 28, and 56 to assess vasomotor and fibrinolytic function. Pulse wave analysis and pulse wave velocity will be measured to assess arterial stiffness on Days -1, 28, and 56.

SECONDARY OUTCOMES:
To investigate the effects of SRT2104 on the reduction of platelet activation markers (platelet-monocyte aggregates). | Serum/plasma/urine research sample(s) will be collected on Days 1, 28, and 56 and will be used to measure platelet activation (platelet-monocyte aggregates).
To evaluate SRT2104 effects on platelet and monocyte surface markers (P-selectin, CD11b), inflammatory markers (high sensitivity CRP, IL-6, SAA, TNF-α and sCD40L), and markers of oxidative stress (urinary and plasma F2-isoprostanes and nitrotyrosine). | Serum/plasma/urine research sample(s) will be collected on Days 1, 28, and 56 to evaluate platelet and monocyte surface markers, inflammatory markers, and markers of oxidative stress.
To characterize the pharmacokinetic profile of SRT2104 after a single dose and multiple administrations in both type 2 diabetes mellitus patients and otherwise healthy smokers in a fed state. | Plasma samples will be collected on Days 1, 28, and 56 at 0h, 15min, 30min, 1, 2, 3, 4, 8, and 12hrs post-dose. Samples will also be collected 24 and 27 hrs post-dose on Days 2, 29, and 57. Also, pre-dose samples will be collected on Days 15 and 43.
To explore the effects of SRT2104 on potential biomarkers of activity for glucose control (HbA1c, glycated albumin and fructosamine) and/or Sirt1 activation. | Serum/plasma/urine research sample(s) will be collected on Days 1, 28, and 56 and will be used to measure potential biomarkers of activity for glucose control.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Noh RM, Venkatasubramanian S, Daga S, Langrish J, Mills NL, Lang NN, Hoffmann E, Waterhouse B, Newby DE, Frier BM. Cardiometabolic effects of a novel SIRT1 activator, SRT2104, in people with type 2 diabetes mellitus. Open Heart. 2017 Sep 2;4(2):e000647. doi: 10.1136/openhrt-2017-000647. eCollection 2017. PMID 28912956
- [Derived] Venkatasubramanian S, Noh RM, Daga S, Langrish JP, Mills NL, Waterhouse BR, Hoffmann E, Jacobson EW, Lang NN, Frier BM, Newby DE. Effects of the small molecule SIRT1 activator, SRT2104 on arterial stiffness in otherwise healthy cigarette smokers and subjects with type 2 diabetes mellitus. Open Heart. 2016 May 17;3(1):e000402. doi: 10.1136/openhrt-2016-000402. eCollection 2016. PMID 27239324
- [Derived] Venkatasubramanian S, Noh RM, Daga S, Langrish JP, Joshi NV, Mills NL, Hoffmann E, Jacobson EW, Vlasuk GP, Waterhouse BR, Lang NN, Newby DE. Cardiovascular effects of a novel SIRT1 activator, SRT2104, in otherwise healthy cigarette smokers. J Am Heart Assoc. 2013 Jun 14;2(3):e000042. doi: 10.1161/JAHA.113.000042. PMID 23770971
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114089 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114089?search=study&search_terms=114089#rs
- Available data/document: Study Protocol: 114089 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114089 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114089 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114089 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114089 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114089 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114089 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register